CLINICAL TRIAL: NCT03313947
Title: Airway Ultrasound to Predict Obstructive Sleep Apnea Syndrome in Children and Its Correlation With Clinical Signs and Symptoms of Obstructive Sleep Apnea
Brief Title: Airway Ultrasound Prediction and Correlation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI was unable to perform ultrasound of airway.
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB17-00436
Record Dates: First submitted 2017-10-16; First posted 2017-10-18 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea; Difficult Airway
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — High-Energy Shock Waves; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Difficult Airway (Other): Ultrasound to measure hyo-mental distance, neutral (Frankfort) position, maximal extended neck position to calculate ratio, width of the tongue between the lingual arteries, and tonsillar size (bilateral).
  Interventions: Procedure: Ultrasound
- Obstructive Sleep Apnea (Other): Ultrasound to measure hyo-mental distance, neutral (Frankfort) position, maximal extended neck position to calculate ratio, width of the tongue between the lingual arteries, and tonsillar size (bilateral).
  Interventions: Procedure: Ultrasound
- Predictive Obstructive Sleep Apnea (Other): The following 6 questions will be asked during the preoperative visit:
  1. While sleeping, does your child snore more than half the time?
  2. While sleeping, does your child always snore?
  3. Have you ever seen your child stop breathing during the night?
  4. Does your child occasionally wet the bed?
  5. Did your child stop growing at a normal rate at any time since birth?
  6. Is your child overweight
  Interventions: Other: Questionnaire

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound to measure hyo-mental distance, neutral (Frankfort) position, maximal extended neck position to calculate ratio, width of the tongue between the lingual arteries, and tonsillar size (bilateral).
  Arms: Difficult Airway; Obstructive Sleep Apnea
Other: Questionnaire — The following 6 questions will be asked during the preoperative visit:
  1. While sleeping, does your child snore more than half the time?
  2. While sleeping, does your child always snore?
  3. Have you ever seen your child stop breathing during the night?
  4. Does your child occasionally wet the bed?
  5. Did your child stop growing at a normal rate at any time since birth?
  6. Is your child overweight
  Arms: Predictive Obstructive Sleep Apnea

SUMMARY:
This is a novel approach to assess the use of ultrasound to support the identification of obstructive sleep apnea syndrome (OSAS) on a screening questionnaire, and potentially to predict a difficult pediatric airway. The investigators hope to determine if a combination of simple bedside clinical tests can be used to identify OSAS in patients who present for surgery with clinical signs of OSAS but without a formal polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* All children presenting for surgery at NCH ranging in age from 3-12 years

Exclusion Criteria:

* Parent/ patient refusal to participate in study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Hyo-mental distance | 5 minutes before surgery starts
  The distance from the hyoid bone to the mentum to predict difficult airway.

SECONDARY OUTCOMES:
Tongue width | 5 minutes after being intubated in surgery
  Width of the tongue between the lingual arteries.
Tonsil size | 5 minutes after being intubated in surgery
  Size of tonsil (bilateral)
Questionnaire | 30 minutes before surgery
  6 predictive OSA questions

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States